CLINICAL TRIAL: NCT00801749
Title: Sleep and Daytime Activity in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nagoya University (Other)
Other Study IDs: 410
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2008-12-08 (Estimated); Status verified 2008-12

CONDITIONS: Cognitive Function
MeSH Terms: interventions — Sleep

INTERVENTIONS:
Behavioral: sleep

SUMMARY:
Sleep relate to cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* patients

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2005-03; Primary Completion 2007-03 (Actual); Study Completion 2008-03 (Actual)